CLINICAL TRIAL: NCT05624970
Title: the Effect of Steady State Aerobic Training on Insulin Sensitivity on Diabetic Patients During Tobacco Cessation
Brief Title: the Effect of Aerobic Training on Insulin Sensitivity on Diabetic Patients During Tobacco Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Naguib Ashry, assistant lecturer at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003343
Record Dates: First submitted 2022-11-10; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Sixty smokers male their age ranged from 40-50 years old will be selected from diabetic outpatient clinic Qasr AL-Einy Hospital. All patients will be carefully examined by the physicians of the hospital. They will be randomly assigned into two groups equal in numbers, as group (A) and group (B).
  Group (A):
  This group will consist of 30 patients who will receive the medical treatment (oral hypoglycemic drugs), aerobic training, tobacco cessation program and nutritional advices for 12 weeks.
  Group (B):
  This group will consist of 30 patients who will receive the medical treatment (oral hypoglycemic drugs), tobacco cessation program and nutritional advices for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) (Experimental): Group (A):
  This group will consist of 30 patients who will receive the medical treatment (oral hypoglycemic drugs), aerobic training, tobacco cessation program and nutritional advices for 12 weeks.
  Interventions: Behavioral: aerobic training , tobacco cessation and nutritional advices
- group (B) (Experimental): Group (B):
  This group will consist of 30 patients who will receive the medical treatment (oral hypoglycemic drugs), tobacco cessation program and nutritional advices for 12 weeks.
  Interventions: Behavioral: tobacco cessation and nutritional advices

INTERVENTIONS:
Behavioral: aerobic training , tobacco cessation and nutritional advices — 1. Aerobic training program according to Taheri et al 2017:
     * Mode: recruits large groups of muscles and includes brisk walking on treadmill, cycling, swimming, and jogging
     * Intensity: submaximal aerobic exercise program (50-60% of maximal heart rate reserve) on treadmill
     * Frequency: 3 sessions a week for 2 months.
     * Duration: 60 min/session The training protocol was divided into three phases: the warm up period (10 minutes), the main program (aerobic exercise; 40 minutes), and a cool down period (10 minutes).
  2. Tobacco Cessation Programs for 3 months
  3. Nutritional advices according to American Diabetes Association (ADA) 2015: for 3 months
  Arms: group (A)
Behavioral: tobacco cessation and nutritional advices — Tobacco Cessation Programs for 3 months Nutritional advices according to American Diabetes Association (ADA) 2015: for 3 months
  Arms: group (B)

SUMMARY:
* Prevalence of smoking in men and women ages 15 and over who currently smoke any tobacco product on a daily or non-daily basis Egypt smoking rate for 2018 was 21.40%, a 0.1% increase from 2016.
* According to WHO reports, smoking is currently responsible for six million premature deaths every year, of which 600 000 individuals die from the effects of second-hand smoke.
* Egypt is one of the 21 countries and territories of the International Diabetes Federation Middle East and North Africa (MENA) region. 463 million people have diabetes in the world and 55 million people in the MENA Region; by 2045 this will rise to 108 million.
* The most profound impact of smoking in diabetic patients is on insulin sensitivity, Cigarette smoking worsens insulin-resistance in patients with diabetes, as smoking decreases subcutaneous absorption of insulin, resulting in increased dosing requirements. When the action of insulin is impaired chronically in smokers, a dose response relationship can be seen between the number of cigarettes smoked and the degree of insulin resistance. Consequently, quitting smoking should improve glycemic control.
* Therefore diabetic patients can get huge benefits from tobacco cessation as they give their bodies chance to decrease percentage of nicotine and increase percentage of insulin so decrease risk of getting atherosclerosis, so smoking cessation improve glycemic control and insulin sensitivity.

DETAILED DESCRIPTION:
Diabetes is a complex, chronic illness requiring continuous medical care with multifactorial risk-reduction strategies beyond glycemic control. Ongoing diabetes self-management education and support are critical to preventing acute complications and reducing the risk of long-term complications.

Nowadays, the harmful effect of smoking is no secret to anyone, unfortunately it is still causes the loss of lives for many adults and young peoples. The Ministry of Health (MOH) seeks to control it and help smokers to quit to save their lives and protect them against smoking-caused diseases such as smoking slows down lung growth in children and teens, increases a person's risk of getting tuberculosis, increases the risk of developing type2 diabetes, also most of COPD (Chronic Obstructive Pulmonary Disease) deaths are a result of smoking. The term "smoking" is not restricted to cigarette smoking only, but includes e-cigarette, shisha and others.

Although cigarette smoking is the leading avoidable cause of death, its specific effects on people with diabetes are even more intricate and profound, thus the macrovascular and microvascular complications become more quickly in smokers with diabetes, and risk of mortality increases. The increased blood pressure and altered lipid profiles in smokers with diabetes could encourage development of the insulin resistance syndrome, setting patients up for further cardiovascular problems.

One of the biggest problems for most patients undergoing a cessation program is the fear of withdrawal symptoms, including cravings, anxiety, depression, irritability, sleep disturbances, increased hunger and weight gain.

Aerobic exercise program for type 2 diabetic has showed great effects not only on glycemic control, blood lipid profiles profile, but also on reducing metabolic risk factors for cardiovascular diseases including insulin resistance. Previous studies have showed the effects of moderate-intensity exercise on the improvement of insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

According to the following:

* All patients will be male.
* Their age between 40-50 years old
* Their BMI 18.5-29.9 kg/m2
* They are diagnosed as type II diabetes for more than 5 years
* Their HbA1c value from > 6.5%
* Smokers for more than10-15 years
* Their smoking index will be moderate and heavy
* All patients are under full medical supervision
* All patients will quit smoking 1-7 days before undergoes aerobic training program

Exclusion Criteria:

All patients will not have:

* Any patient is known to have any unstable medical condition.
* Any musculoskeletal or neurological disorder
* Hepatic diseases.
* Kidney disorders
* Type I diabetes mellitus
* Type II insulin
* Uncontrolled hypertension
* Unstable angina pectoris
* Uncompensated heart failure
* Recent myocardial infarction
* Heart block
* Cerebrovascular disease
* Anemia
* Patients whose smoking index light
* Tobacco smokers less than 20 years

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | 3 months
  The Homeostasis Model Assessment (HOMA):
  HOMA-IR = [(Fasting Insulin (µU/mL)) X (Fasting Glucose (mmol/L))]/22.5

SECONDARY OUTCOMES:
assessment of glycemic control | 3 months
  HbA1c
blood pressure | 3 months
  Normal blood pressure: systolic < 140 mmHg, diastolic <90 mmHg
heart rate | 3 months
  Normal resting heart rate 60-90 beats per minute
respiratory rate | 3 months
  Normal respiratory rate for healthy adults is between 12 and 20 breaths per minute.
oxygen saturation | 3 months
  A pulse oximeter can measure oxygen saturation. The generally accepted standard is that a normal resting oxygen saturation of less than 95% is considered abnormal
ankle brachial index | 3 months
  The ankle-brachial index (ABI) is the ratio of the systolic blood pressure (SBP) measured at the ankle to that measured at the brachial artery, it was shown that the ABI is an indicator of atherosclerosis and peripheral arterial disease(PAD) The ABI threshold most commonly used is ≤0.90.
smoking abstintent questionnaire | 3 months
  The Smoking Abstinence Questionnaire, appears to capture reliably smokers' expectancies for abstinence (Withdrawal, Social Improvement/Non-smoker Identity, Adverse Outcomes, Common Reasons, Optimistic Outcomes, Coffee Use, and Weight Gain) and expectancies related to the success of a quit attempt (Treatment Effectiveness, Barriers to Treatment and Social Support). It remains to be seen how far any of these expectancies predict attempts to quit, withdrawal, treatment utilization and response and quitting success above and beyond existing measures.
smoking index | 3 months
  cigarette per day multiplied by years of smoking
A body shape index (ABSI) | 3 months
  WC divided by (BMI 2/3 multiplied by height 1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Elnahas, professor, Study Director — Cairo Univeristy; Rana elbanaa, lecturer, Study Director — Cairo Univeristy; Yasmine mohamed, lectuere, Study Director — cairo univeristy
Locations (1):
- Alaa mohamed Naguib, Cairo, Egypt